CLINICAL TRIAL: NCT06222788
Title: Breast Cancer Plasma Adjuvant Intra-operative Treatment (Breast Cancer PAINT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Ozmosis Research Inc. (Industry); Ministère de l'Économie, de l'Innovation et de l'Énergie, Québec, Canada (Unknown); Quebec Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-11512; OZM-133 (Other: Ozmosis Research Inc.)
Record Dates: First submitted 2023-12-13; First posted 2024-01-25 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: non-thermal plasma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NTP treatment (Experimental): The patients will be treated with NTP intra-operatively.
  Interventions: Device: Convertible Plasma Jet

INTERVENTIONS:
Device: Convertible Plasma Jet — NTP will be applied to the patients using the Convertible Plasma Jet (CPJ, NexPlasmaGen Inc.)

SUMMARY:
The goal of this clinical trial is to test the safety of the use of non-thermal plasma (NTP, an ionized gas) on the tumor bed after the removal of the tumor in breast cancer patients. The main questions it aims to answer are:

* To determine the safe and tolerable dose of NTP in patients with breast cancer;
* To assess the safety and tolerability of NTP;
* To assess the cosmetic effects of NTP treatment in patients with breast cancer. Participants will receive one treatment of the tumor bed after the removal of their breast tumor.

DETAILED DESCRIPTION:
Non-thermal plasma (NTP) refers to an ionized gas composed of ions, electrons and other reactive agents. The anti-cancerous properties of NTP have been proven in vitro and in vivo. The 10-year local recurrence risk (LRR) in breast cancer patients after a breast conservation therapy (i.e., lumpectomy, typically followed by radiation therapy) is still as high as 15-20%. NTP could be used to further treat the tumor bed to reduce the LRR.

The primary objective of this clinical trial is to determine the safe and tolerable dose of NTP treatment following breast cancer lumpectomy. The secondary objectives are to assess the safety and tolerability of NTP and to assess the cosmetic effects of NTP treatment in patients with breast cancer. Our exploratory objective is to assess the impact of NTP treatment on cancerous and normal tissues. Patients are followed for 3 months after NTP treatment. The patients are divided into 3 groups: group A (n=3): NTP treatment of part of the tumor bed ex vivo. Group B (n=3): NTP treatment of part of the tumor bed in situ (all treated tissues are removed for analysis). Group C (n=6-24): dose escalation per "3+3 Design" up to a maximum dose level 3. NTP treatment of part of the tumor bed in situ (the treated parts of the tumor bed will not be excised, except a small portion for analysis).

The safety and tolerability of treatment will be evaluated by means of dose limiting toxicities, adverse events (AEs) and serious adverse events reports, physical examinations, and laboratory safety evaluations. AEs will be coded according to the CTCAE v5.0. The results will be tabulated to examine their frequency, grade, and relationship to study treatment. The results of laboratory assessments will be evaluated similarly. The number of patients with cosmetic alterations linked to the NTP treatment and type of alterations will be assessed through the quality of life questionnaires (questions on breast appearance and texture) and through the photo collection. This is the first clinical trail to study the safety and tolerability of NTP in an all breast-cancer patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing study consent.
2. ECOG ≤2.
3. Patient with T1-4 breast cancer for groups A and B; patient with T1/T2 breast cancer for group C (based on physical exam, not radiological measurements).
4. Patient is scheduled to undergo a lumpectomy.

Exclusion Criteria:

1. Prior treatment for the tumor of interest (including chemotherapy, immunotherapy, radiotherapy).
2. Patient planning to or undergoing intraoperative radiotherapy.
3. Diabetes (types I and II).
4. Hypercortisolism.
5. Collagen vascular disease.
6. Patient requiring systemic corticosteroids at physiologic doses exceeding 10 mg/day of prednisone or its equivalent.
7. Patient receiving daily chemotherapy for rheumatological conditions.
8. Pregnancy (a urine pregnancy test must be obtained for non-sterile women of childbearing potential prior to surgery).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incremental increase of NTP dose to reach maximum safe dose. | 3 months
  The safety and tolerability of treatment will be evaluated by means of dose-limiting toxicities, adverse events and serious adverse events reports, physical examinations, and laboratory safety evaluations. Dose-limiting toxicities are defined as a grade 4 fever, breast infection, skin ulceration or chest wall necrosis (according to CTCAE v5.0).

SECONDARY OUTCOMES:
Number of patients with adverse events linked to the NTP treatment and type of events. | 3 months
  Adverse events will be coded according to the CTCAE Version 5.0. The results will be tabulated to examine their frequency, organ systems affected, grade, and relationship to study treatment.
Number of patients with cosmetic alterations linked to the NTP treatment and type of alterations. | 3 months
  This will be assessed through the quality of life questionnaires (questions on breast appearance and texture) and through the photo collection (pictures of the treated breast before/after NTP treatment).

OTHER OUTCOMES:
Evidence of cancer cell death and effects on normal tissue in samples treated with NTP ex vivo or in situ. | 15 months
  Ex vivo or in situ treatment of cancerous and normal tissues with NTP followed by fixation of the tissues and analysis by immunofluorescence.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal - CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glory A, Patocskai E, Wong P. Breast cancer PAINT: a first-in-human, dose-escalation study to determine the safety of Plasma Adjuvant INtra-operative Treatment in breast cancer patients. BMC Cancer. 2025 Apr 22;25(1):748. doi: 10.1186/s12885-025-14153-5. PMID 40264065